CLINICAL TRIAL: NCT03424876
Title: A Retrospective Cohort Study
Brief Title: To Compare the Efficacy of Surgery Followed by Sunitinib With Surgery Followed by Imatinib in GIST Patients With Progression on Imatinib.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Shen Lin, Professor, Peking University
Other Study IDs: G0602
Record Dates: First submitted 2018-01-03; First posted 2018-02-07 (Actual); Last update posted 2018-03-01 (Actual); Status verified 2018-02

CONDITIONS: GIST
Keywords: Sunitinib Imatinib
MeSH Terms: interventions — Imatinib Mesylate; Sunitinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Gene c-kit/PDGFRA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Arm A: Imatinib 400 mg/day or 600mg/day, and within 6 weeks after surgery, continuous treatment was not tolerated until tumor progression, recurrence or adverse reactions were not tolerated.
  Interventions: Drug: Imatinib 400mg
- Arm B: Sunitinib 37.5 mg/day, continuous taking, or 50 mg/day (4/2), began within 6 weeks after surgery, and was continuously administered until tumor progression, recurrence or adverse reactions were not tolerated
  Interventions: Drug: Sunitinib 37.5Mg Oral Capsule

INTERVENTIONS:
Drug: Imatinib 400mg — exposure 400 mg/day or 600mg/day,
  Groups: Arm A
Drug: Sunitinib 37.5Mg Oral Capsule — exposure 37.5 mg/day, continuous taking, or 50 mg/day (4/2)
  Groups: Arm B

SUMMARY:
To compare the efficacy of surgery followed by sunitinib with surgery followed by imatinib in GIST patients with progression on imatinib;To investigate the optimal therapy after surgery in GIST patients with focal or multifocal progression in imatinib

DETAILED DESCRIPTION:
Primary Endpoint: To evaluate the progression free survival of the patients with progression receiving surgery followed by sunitinib therapy comparing with surgery followed by imatinib Secondary Endpoint：To evaluate the overall survival of the patients with progression receiving surgery followed by sunitinib therapy comparing with surgery followed by imatinib the relationship of c-kit secondary mutation and progression free survival of surgery followed by TKI therapy the safety and tolerability of the two therapy.

Statistics:All the statistical analysis is performed using SPSS version 20.0 (IBM corporation, United States). Pearson's chi-squared test was used to compare categorical variables. PFS and OS analyses were estimated with Kaplan-Meier method and log-rank test and multivariable analyses were performed to assess survival difference. A two sided p-value of <0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

1. .Histopathological diagnosis of metastatic GIST.
2. . After the treatment of imatinib, imatinib 400mg/day after treatment, the tumor generalized.
3. . Patients with generalized progress were satisfied with tumor reduction after imatinib resistance for various reasons.
4. at least 1 month after surgery for imatinib treatment or sunitinib treatment.
5. at least one imaging assessment was received after surgery.
6. . Complete clinical data and follow-up data.

Exclusion Criteria:

1. . Before operation, he was treated with sunitinib
2. . Patients receiving tumor reduction were not satisfied with the standard of the reduction of tumor.
3. . The treatment of imatinib or sunitinib after surgery was less than 1 month.
4. . Incomplete clinical data or follow-up data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Test group is imatinib 400 mg/day or higher dose treatment failure and satisfactory reduction of tumor surgery patients with advanced gastrointestinal stromal tumor, patients must meet all the inclusion criteria and exclusion criteria to enter test.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2017-06-02 (Actual); Primary Completion 2018-06-02 (Estimated); Study Completion 2018-08-08 (Estimated)

PRIMARY OUTCOMES:
Efficiency | 12 months
  The curative effect was evaluated by measuring the unprogression-survival (PFS) each treatment group.
Security | 12 months
  Clinical and laboratory toxicity/symptoms will be graded according to the nci-ctc toxicity criteria.
Molecular marker detection | 12 months
  Gene mutation of c-kit/PDGFRA of imatinib resistance

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided
IPD will be shared later

REFERENCES:
- [Background] Abrams TJ, Lee LB, Murray LJ, Pryer NK, Cherrington JM. SU11248 inhibits KIT and platelet-derived growth factor receptor beta in preclinical models of human small cell lung cancer. Mol Cancer Ther. 2003 May;2(5):471-8. PMID 12748309
- [Background] Rubin BP, Singer S, Tsao C, Duensing A, Lux ML, Ruiz R, Hibbard MK, Chen CJ, Xiao S, Tuveson DA, Demetri GD, Fletcher CD, Fletcher JA. KIT activation is a ubiquitous feature of gastrointestinal stromal tumors. Cancer Res. 2001 Nov 15;61(22):8118-21. PMID 11719439
- [Background] Li J, Gao J, Hong J, Shen L. Efficacy and safety of sunitinib in Chinese patients with imatinib-resistant or -intolerant gastrointestinal stromal tumors. Future Oncol. 2012 May;8(5):617-24. doi: 10.2217/fon.12.29. PMID 22646775
- [Result] Fletcher CD, Berman JJ, Corless C, Gorstein F, Lasota J, Longley BJ, Miettinen M, O'Leary TJ, Remotti H, Rubin BP, Shmookler B, Sobin LH, Weiss SW. Diagnosis of gastrointestinal stromal tumors: A consensus approach. Hum Pathol. 2002 May;33(5):459-65. doi: 10.1053/hupa.2002.123545. PMID 12094370
- [Result] Blackstein ME, Blay JY, Corless C, Driman DK, Riddell R, Soulieres D, Swallow CJ, Verma S; Canadian Advisory Committee on GIST. Gastrointestinal stromal tumours: consensus statement on diagnosis and treatment. Can J Gastroenterol. 2006 Mar;20(3):157-63. doi: 10.1155/2006/434761. PMID 16550259
- [Result] Goettsch WG, Bos SD, Breekveldt-Postma N, Casparie M, Herings RM, Hogendoorn PC. Incidence of gastrointestinal stromal tumours is underestimated: results of a nation-wide study. Eur J Cancer. 2005 Dec;41(18):2868-72. doi: 10.1016/j.ejca.2005.09.009. Epub 2005 Nov 15. PMID 16293410
- [Result] DeMatteo RP, Lewis JJ, Leung D, Mudan SS, Woodruff JM, Brennan MF. Two hundred gastrointestinal stromal tumors: recurrence patterns and prognostic factors for survival. Ann Surg. 2000 Jan;231(1):51-8. doi: 10.1097/00000658-200001000-00008. PMID 10636102
- [Result] Graadt van Roggen JF, van Velthuysen ML, Hogendoorn PC. The histopathological differential diagnosis of gastrointestinal stromal tumours. J Clin Pathol. 2001 Feb;54(2):96-102. doi: 10.1136/jcp.54.2.96. PMID 11215292
- [Result] Mendel DB, Laird AD, Xin X, Louie SG, Christensen JG, Li G, Schreck RE, Abrams TJ, Ngai TJ, Lee LB, Murray LJ, Carver J, Chan E, Moss KG, Haznedar JO, Sukbuntherng J, Blake RA, Sun L, Tang C, Miller T, Shirazian S, McMahon G, Cherrington JM. In vivo antitumor activity of SU11248, a novel tyrosine kinase inhibitor targeting vascular endothelial growth factor and platelet-derived growth factor receptors: determination of a pharmacokinetic/pharmacodynamic relationship. Clin Cancer Res. 2003 Jan;9(1):327-37. PMID 12538485
- [Result] O'Farrell AM, Abrams TJ, Yuen HA, Ngai TJ, Louie SG, Yee KW, Wong LM, Hong W, Lee LB, Town A, Smolich BD, Manning WC, Murray LJ, Heinrich MC, Cherrington JM. SU11248 is a novel FLT3 tyrosine kinase inhibitor with potent activity in vitro and in vivo. Blood. 2003 May 1;101(9):3597-605. doi: 10.1182/blood-2002-07-2307. Epub 2003 Jan 16. PMID 12531805
- [Result] Schlessinger J. Cell signaling by receptor tyrosine kinases. Cell. 2000 Oct 13;103(2):211-25. doi: 10.1016/s0092-8674(00)00114-8. No abstract available. PMID 11057895
- [Result] Bello C. B. Houk, L. Sherman, et al. Effect of rifampin on the pharmacokinetics of SU11248 in healthy volunteers. Proc.ASCO abstr#3078, 2005.
- [Result] Blanke CD, Rankin C, Demetri GD, Ryan CW, von Mehren M, Benjamin RS, Raymond AK, Bramwell VH, Baker LH, Maki RG, Tanaka M, Hecht JR, Heinrich MC, Fletcher CD, Crowley JJ, Borden EC. Phase III randomized, intergroup trial assessing imatinib mesylate at two dose levels in patients with unresectable or metastatic gastrointestinal stromal tumors expressing the kit receptor tyrosine kinase: S0033. J Clin Oncol. 2008 Feb 1;26(4):626-32. doi: 10.1200/JCO.2007.13.4452. PMID 18235122
- [Result] Zalcberg JR, Verweij J, Casali PG, Le Cesne A, Reichardt P, Blay JY, Schlemmer M, Van Glabbeke M, Brown M, Judson IR; EORTC Soft Tissue and Bone Sarcoma Group, the Italian Sarcoma Group; Australasian Gastrointestinal Trials Group. Outcome of patients with advanced gastro-intestinal stromal tumours crossing over to a daily imatinib dose of 800 mg after progression on 400 mg. Eur J Cancer. 2005 Aug;41(12):1751-7. doi: 10.1016/j.ejca.2005.04.034. PMID 16098458
- [Result] Demetri GD, van Oosterom AT, Garrett CR, Blackstein ME, Shah MH, Verweij J, McArthur G, Judson IR, Heinrich MC, Morgan JA, Desai J, Fletcher CD, George S, Bello CL, Huang X, Baum CM, Casali PG. Efficacy and safety of sunitinib in patients with advanced gastrointestinal stromal tumour after failure of imatinib: a randomised controlled trial. Lancet. 2006 Oct 14;368(9544):1329-38. doi: 10.1016/S0140-6736(06)69446-4. PMID 17046465
- [Result] Demetri GD, Garrett CR, Schoffski P, Shah MH, Verweij J, Leyvraz S, Hurwitz HI, Pousa AL, Le Cesne A, Goldstein D, Paz-Ares L, Blay JY, McArthur GA, Xu QC, Huang X, Harmon CS, Tassell V, Cohen DP, Casali PG. Complete longitudinal analyses of the randomized, placebo-controlled, phase III trial of sunitinib in patients with gastrointestinal stromal tumor following imatinib failure. Clin Cancer Res. 2012 Jun 1;18(11):3170-9. doi: 10.1158/1078-0432.CCR-11-3005. PMID 22661587
- [Result] Vincenzi B, Nannini M, Fumagalli E, Bronte G, Frezza AM, De Lisi D, Spalato Ceruso M, Santini D, Badalamenti G, Pantaleo MA, Russo A, Dei Tos AP, Casali P, Tonini G. Imatinib dose escalation versus sunitinib as a second line treatment in KIT exon 11 mutated GIST: a retrospective analysis. Oncotarget. 2016 Oct 25;7(43):69412-69419. doi: 10.18632/oncotarget.5136. PMID 26416414
- [Result] Hsu CC, Wu CE, Chen JS, Tseng JH, Chiang KC, Liu YY, Tsai CY, Cheng CT, Chen TW, Jan YY, Yeh TS, Chen YY, Yeh CN. Imatinib escalation or sunitinib treatment after first-line imatinib in metastatic gastrointestinal stromal tumor patients. Anticancer Res. 2014 Sep;34(9):5029-36. PMID 25202087
- [Result] Fairweather M, Balachandran VP, Li GZ, Bertagnolli MM, Antonescu C, Tap W, Singer S, DeMatteo RP, Raut CP. Cytoreductive Surgery for Metastatic Gastrointestinal Stromal Tumors Treated With Tyrosine Kinase Inhibitors: A 2-institutional Analysis. Ann Surg. 2018 Aug;268(2):296-302. doi: 10.1097/SLA.0000000000002281. PMID 28448384
- [Result] Raut CP, Posner M, Desai J, Morgan JA, George S, Zahrieh D, Fletcher CD, Demetri GD, Bertagnolli MM. Surgical management of advanced gastrointestinal stromal tumors after treatment with targeted systemic therapy using kinase inhibitors. J Clin Oncol. 2006 May 20;24(15):2325-31. doi: 10.1200/JCO.2005.05.3439. PMID 16710031
- [Result] DeMatteo RP, Maki RG, Singer S, Gonen M, Brennan MF, Antonescu CR. Results of tyrosine kinase inhibitor therapy followed by surgical resection for metastatic gastrointestinal stromal tumor. Ann Surg. 2007 Mar;245(3):347-52. doi: 10.1097/01.sla.0000236630.93587.59. PMID 17435539
- [Result] Gronchi A, Fiore M, Miselli F, Lagonigro MS, Coco P, Messina A, Pilotti S, Casali PG. Surgery of residual disease following molecular-targeted therapy with imatinib mesylate in advanced/metastatic GIST. Ann Surg. 2007 Mar;245(3):341-6. doi: 10.1097/01.sla.0000242710.36384.1b. PMID 17435538